CLINICAL TRIAL: NCT03540524
Title: Assessment of Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Multiple Oral Doses of the Combination of GLPG2451 and GLPG2222, With or Without GLPG2737, in Adult Subjects With Cystic Fibrosis
Brief Title: A Study Looking at the Safety, Tolerability and Efficacy of the Combination of the Study Drugs GLPG2451 and GLPG2222 With or Without GLPG2737 in Patients With Cystic Fibrosis.
Acronym: FALCON
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLPG2737-CL-105; 2017-001067-20 (EudraCT Number)
Record Dates: First submitted 2018-04-27; First posted 2018-05-30 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2018-04

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — GLPG2222

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A - F508del homozygous (Experimental): Dual combination (GLPG2451 and GLPG2222) will be administered for 14 days, followed by the triple combination (GLPG2451, GLPG2222 and GLPG2737) for 14 days, without washout in between the sequential treatment periods.( Study Part I)
  Interventions: Drug: GLPG2451 dose regimen A; Drug: GLPG2222; Drug: GLPG2737
- Cohort B - F508del heterozygous/potentiator nonresponsive (Experimental): Dual combination (GLPG2451 and GLPG2222) will be administered for 14 days, followed by the triple combination (GLPG2451, GLPG2222 and GLPG2737) for 14 days, without washout in between the sequential treatment periods. (study Part II)
  Interventions: Drug: GLPG2451 dose regimen B; Drug: GLPG2222; Drug: GLPG2737
- Cohort C - F508del homozygous (Experimental): Dual combination (GLPG2451 and GLPG2222) will be administered for 14 days, followed by the triple combination (GLPG2451, GLPG2222 and GLPG2737) for 14 days, without washout in between the sequential treatment periods. (Study Part II)
  Interventions: Drug: GLPG2451 dose regimen B; Drug: GLPG2222; Drug: GLPG2737

INTERVENTIONS:
Drug: GLPG2451 dose regimen A — GLPG2451 oral suspension, daily.
  Arms: Cohort A - F508del homozygous
Drug: GLPG2451 dose regimen B — GLPG2451 oral suspension, daily.
  Arms: Cohort B - F508del heterozygous/potentiator nonresponsive; Cohort C - F508del homozygous
Drug: GLPG2222 — GLPG2222 tablet for oral use, daily.
Drug: GLPG2737 — GLPG2737 capsules for oral use, daily.

SUMMARY:
This is a Phase Ib, multi-center, open-label, nonrandomized multiple cohorts study to assess the safety, tolerability, pharmacokinetics, and pharmacodynamics of multiple doses of a combination treatment of GLPG2451 and GLPG2222, with and without GLPG2737, in adult subjects with Cystic Fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Female or male subject ≥18 years of age, on the day of signing the Informed Consent Form (ICF)
* Confirmed clinical diagnosis of cystic fibrosis (CF) (documented in the subject's medical record).
* Eligible cystic fibrosis transmembrane conductance regulator (CFTR) genotype at screening:

  * Cohort A: Homozygous for the F508del CFTR mutation
  * Cohort B: Heterozygous for the F508del CFTR mutation with a potentiator non-responsive mutation on the second allele
  * Cohort C: Homozygous for the F508del CFTR mutation
* A body weight of ≥40 kg at screening.
* Stable concomitant medication for pulmonary health for CF for at least 4 weeks prior to the first study drug administration and planned continuation of the same concomitant medication for the duration of the dosing period of the study. Subjects with diabetes mellitus and/or pancreatic insufficiency are eligible for the study provided they are on stable treatment (e.g. medication, diet, pancreatic enzyme replacement therapy) for at least 4 weeks prior to the first study drug administration in the opinion of the investigator.
* Forced expiratory volume in 1 second (FEV1): 40% ≤ FEV1 ≤ 90% of predicted normal for age, sex, and height at screening (pre- or post bronchodilator) at screening.
* Sweat chloride concentration ≥60 mmol/L at screening.
* Non-smoker and non-user of any nicotine and or cannabis containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to the screening. A non-user is defined as an individual who has abstained from any nicotine containing products for at least 1 year prior to the screening.

Exclusion Criteria:

* History of or ongoing allergic bronchopulmonary aspergillosis.
* Medical history of cataract (or lens opacity) and/or glaucoma.
* Cataract (or lens opacity) and/or glaucoma determined by an ophthalmologist during the screening period.
* Unstable pulmonary status or respiratory tract infection (including rhinosinusitis) requiring a change in therapy within 4 weeks prior to the first study drug administration.
* History of clinically meaningful unstable or uncontrolled chronic disease that makes the subject unsuitable for inclusion in the study in the opinion of the investigator.
* Need for supplemental oxygen during the day, and >2 L/minute while sleeping.
* History of hepatic cirrhosis with portal hypertension (e.g., signs/symptoms of splenomegaly, esophageal varices).
* History of malignancy within the past 5 years (except for basal cell carcinoma of the skin with no evidence of recurrence and/or carcinoma in situ of the cervix that has been treated with no evidence of recurrence).
* Use of any moderate and strong inhibitor(s) or inducer(s) of CYP3A4 within 4 weeks prior to the first study drug administration (e.g., clarithromycin, itraconazole, ketoconazole, telithromycin, rifampin, carbamazepine).
* Use of CFTR modulator therapy (e.g., lumacaftor and/or ivacaftor) within 4 weeks prior to the first study drug administration.
* Use of any oral corticosteroid within 3 months of screening; or history of oral corticosteroid use for ≥30 days (cumulative) within 2 years of screening.
* Abnormal liver function test at screening; defined as aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) and/or alkaline phosphatase and/or gamma-glutamyl transferase (GGT) ≥3× the upper limit of normal (ULN); and/or total bilirubin ≥1.5× the ULN.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-31 (Actual); Primary Completion 2019-03-11 (Actual); Study Completion 2019-03-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with adverse events. | Up to 24 weeks after the last dose
  To assess safety and tolerability of doses of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I and Part II).
Maximum observed plasma concentration (Cmax). | Day 14
  To characterize the pharmacokinetics (PK) of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).
Maximum observed plasma concentration (Cmax). | Day 28
  To characterize the PK of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).
Area under the plasma concentration-time curve from time zero until 24 hours (AUC0-24h). | Day 14
  To characterize the PK of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).
Area under the plasma concentration-time curve from time zero until 24 hours (AUC0-24h). | Day 28
  To characterize the PK of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).
Trough plasma concentration observed at the end of the dosing interval (24 hours post-dose) (Ctrough). | Between Day 2 and Day 28
  To characterize the PK of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I and Part II).
Change from baseline in sweat chloride concentration. | Between Day 1 pre-dose and Day 28
  To assess changes in sweat chloride concentration after administration of the combination of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part II).
Change from baseline in percent predicted FEV1. | Between Day 1 pre-dose and Day 28
  To assess changes in percent predicted FEV1 after administration of the combination of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part II).

SECONDARY OUTCOMES:
Change from baseline in sweat chloride concentration. | Between Day 1 pre-dose and Day 28
  To assess changes in sweat chloride concentration after administration of the combination of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).
Change from baseline in percent predicted FEV1. | Between Day 1 pre-dose and Day 28
  To assess changes in percent predicted FEV1 after administration of the combination of GLPG2451 and GLPG2222 with or without GLPG2737 (Study Part I).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Van de Steen, MD MBA, Study Director — Galapagos NV
Locations (20):
- Belgium (4):
  - Study Site BEL004, Antwerp
  - Study Site BEL003, Brussels
  - Study Site BEL002, Ghent
  - Study Site BEL001, Leuven
- Study Site BGR001, Sofia, Bulgaria
- Germany (2):
  - Study Site DEU001, Berlin
  - Study Site DEU002, Essen
- Study Site GRC001, Thessaloniki, Greece
- Netherlands (2):
  - Study Site NLD002, Amsterdam
  - Study Site NLD001, Utrecht
- Study Site SRB001, Belgrade, Serbia
- Sweden (2):
  - Study Site SWE001, Gothenburg
  - Study Site SWE002, Stockholm
- United Kingdom (7):
  - Study Site GBR003, Birmingham
  - Study Site GBR004, Glasgow
  - Study Site GBR005, Liverpool
  - Study Site GBR007, London
  - Study Site GBR006, Newcastle
  - Study Site GBR001, Papworth Everard
  - Study Site GBR002, Wythenshawe